CLINICAL TRIAL: NCT03110328
Title: Phase II Study of Pembrolizumab in Metastatic Biliary Tract Cancer as Second-line Treatment After Failing to at Least One Cytotoxic Chemotherapy Regimen: Integration of Genomic Analysis to Identify Predictive Molecular Subtypes
Brief Title: Study of Pembrolizumab in Metastatic Biliary Tract Cancer as Second-line Treatment After Failing to at Least One Cytotoxic Chemotherapy Regimen: Integration of Genomic Analysis to Identify Predictive Molecular Subtypes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seung tae Kim,PhMD, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-12-145
Record Dates: First submitted 2017-03-16; First posted 2017-04-12 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Pembrolizumab (MK-3475) 200 mg every 3 weeks (Q3W)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mk3475 200mg (Experimental): Pembrolizumab (MK-3475) 200 mg every 3 weeks (Q3W) Open-label
  Interventions: Drug: MK3475

INTERVENTIONS:
Drug: MK3475 — anti-PD1 immunotherapy
  Other Names: Pembrolizumab

SUMMARY:
eligible subjects will receive treatment beginning on Day 1 of each 3-week dosing cycle for pembrolizumab. Treatment with pembrolizumab will continue until documented disease progression, unacceptable adverse event(s),intercurrent illness that prevents further administration of treatment, Investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, subject receives 24 months of pembrolizumab, or administrative reasons requiring cessation of treatment.

DETAILED DESCRIPTION:
This is a single-arm, single-center, open-label trial of pembrolizumab (MK-3475) in subjects with metastatic biliary tract cancer as second-line treatment after failing to at least one cytotoxic chemotherapy regimen

Approximately 33 subjects will be enrollment to evaluate the efficacy and safety of pembrolizumab.

Enrollment will begin with all subjects without regard for PD-L1 expression status.

An evaluable specimen for PD-L1 status must be available and confirmed prior to enrollment.

All study subjects will be evaluated every 6 weeks (+/- 7 days) following the date of IP drug adminstration for the first six months and every 12 weeks (+/- 7 days) thereafter until progression of disease is documented with radiologic imaging (computed tomography or magnetic resonance imaging).

The primary efficacy endpoint is ORR (objective response rate) per RECIST 1.1. If a subject has progression of disease by RECIST 1.1, it is recommended that the subject be discontinued from the study treatment unless, in the Investigator's opinion, the subject is deriving benefit from treatment.

Adverse events will be monitored throughout the trial and graded in severity according to the guidelines outlined in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

Except as noted above, treatment with pembrolizumab will continue until documented disease progression, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, Investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, completion of 24 months of pembrolizumab, or administrative reasons requiring the cessation of treatment.

After the end of treatment, each subject will be followed for 30 days for adverse event monitoring (serious adverse events and events of clinical interest will be collected for 90 days after the end of treatment or 30 days after the end of treatment if the subject initiates new anticancer therapy, whichever is earlier).Subjects who discontinue treatment for reasons other than disease progression will have post-treatment follow-up for disease status until disease progression, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up. All subjects will be followed by telephone contact for overall survival until death, withdrawal of consent or the end of the study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically-confirmed diagnosis of biliary tract cancer including intra- and extra-hepatic biliary tract cancer
2. Have metastatic disease or locally advanced, unresectable disease with feasible biopsy sites (baseline and follow up)
3. Has experienced documented objective radiographic or clinical disease progression during or after first-line therapy containing any platinum/gemcitabine or any platinum/ fluoropyrimidine doublet.
4. Have measurable disease based on RECIST as determined by investigator. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
5. Be willing to provide fresh tissue for biomarker analysis, and, based on the adequacy of the tissue sample quality for assessment of biomarker status. Repeat samples may be required if adequate tissue is not provided. Newly obtained endoscopic biopsy specimens are preferred to archived samples and formalin-fixed, paraffin-embedded (FFPE) block specimens are preferred to slides.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has squamous cell or sarcomatoid biliary duct cancer. Ampulla of Vater cancer. Gall bladder cancer
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has a known history of active TB (Bacillus Tuberculosis)
5. Hypersensitivity to pembrolizumab or any of its excipients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Best overall response | 12months
  Integrative genomic analysis to identify association of response and OS) and primary resistance to pembrolizumab with key genomic markers for immunotherapy
progression-free survival | 12months
  Integrative genomic analysis to identify association of response and OS) and primary resistance to pembrolizumab with key genomic markers for immunotherapy
overall survival | 12months
  Integrative genomic analysis to identify association of response and OS) and primary resistance to pembrolizumab with key genomic markers for immunotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea